CLINICAL TRIAL: NCT00530725
Title: Prospective Randomized Trial of the Management of Occult Pneumothoraces in Mechanically Ventilated Patients
Brief Title: Management of Occult Pneumothoraces in Mechanically Ventilated Patients
Acronym: OPTICC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: CHU de Quebec-Universite Laval (Other); Sunnybrook Health Sciences Centre (Other); Canadian Intensive Care Foundation (Other); London Health Sciences Centre (Other); Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Andrew W Kirkpatrick, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPTICC Trial
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Pneumothorax
Keywords: occult pneumothorax; mechanical ventilation; critical care; pneumothorax; thoracostomy
MeSH Terms: conditions — Pneumothorax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- chest drainage (Active Comparator): This represents the best current standard of care although this is quite controversial
  Interventions: Procedure: chest drainage
- close observation (Experimental): This is the novel approach that has some justification in the literature
  Interventions: Other: close clinical observation

INTERVENTIONS:
Procedure: chest drainage — may be a chest tube of chest drainage procedure of any type (ie formal tube, pig-tail catheter, etc)
  Arms: chest drainage
Other: close clinical observation — close clinical observation in an operating room or intensive care unit without active intervention
  Arms: close observation

SUMMARY:
Collapsed lungs are common injuries after traumatic injury that regularly cause needless deaths despite being treatable with chest tubes. Properly used these tubes can be life-saving. Unfortunately, improperly used they can cause pain, bleeding, and other fatal complications themselves. Over the last few decades with increased use of CT scanning it is apparent that many small collapsed lungs are not seen on chest X-rays, and there is little guidance for the treating Doctors as to how to treat these patients. There is almost no good data that tells us whether these smaller pneumothoraces require treatment with chest tubes or whether they can simply be closely watched. This proposal is to carry out a simple trial of randomly assigning patients who do not appear to have any symptoms or problems from their occult pneumothorax to either having a standard chest tube or to being watched. Our careful review of the medical literature indicates that the investigators cannot honestly tell patients and their families which treatment is best or required. Our audit of current practice also indicates that Doctors in Calgary and across Canada, regularly prescribe both treatments regularly but in a hap-hazard. The patients in this study will be very closely watched in the intensive care unit and if they develop any breathing problems and do not have a chest tube in, then one will be inserted. The main results that the investigators are trying to determine with this pilot study, though, is whether the investigators are able to detect appropriate patients, to recruit them into such a study, and whether the guidelines the investigators have created to manage these patients in this study will be acceptable to all the patient's care givers. This data will help us to design a future large multi-centre trial that will hopefully provide information as how best to manage this type of injured patient.

DETAILED DESCRIPTION:
The term "Occult Pneumothorax" (OPTX), describes a pneumothorax (PTX) that while not suspected on the basis of either clinical examination or plain radiograph, is ultimately detected with thoraco-abdominal computed tomograms (CT). This situation is increasingly common in contemporary trauma care with the increased use of CT. The incidence appears to approximately 5% in injured populations presenting to hospital, with CT revealing at least twice as many PTXs as suspected on plain radiographs. While PTXs are a common and treatable (through chest drainage) cause of mortality and morbidity, there is clinical equipoise and significant disagreement regarding the appropriate treatment of the OPTX. Based on level III evidence, some authors have recommended observation without chest drainage for all but the largest OPTXs, recommendations that contravene the standard dictum for ventilated patients as recommended by the Advanced Trauma Life Support Course of the American College of Surgeons. The controversy is the greatest in the critical care unit population who require positive pressure ventilation. This is also the group for whom the highest rates of chest tube complications have been reported. Complication rates related to chest tubes in general, have been claimed in up to 21% of cases.

No previous studies have focused specifically on the population of mechanically ventilated patients. There have been only 45 reported ventilated trauma patients ever randomized to treatment or observation. Enderson found that 8 (53%) of 15 patients had PTX progression with 3 tension pneumothoraces. Brasel found that of 9 observed OPTXs, 2 progressed. Brasel concluded observation was safe, while Enderson felt chest tubes were mandatory. The investigators thus propose to carry out a prospective randomized trial to examine the need for chest drainage in small to moderate sized OPTX's, as well as the practicalities of carrying out such a study.

The experience and knowledge gained from this pilot will be intended to provide additional support to a future submission to the Canadian Institute for Health Research in order to carry out a multi-centre prospective trial involving the member institutions of the Canadian Trauma Trials Collaborative (CTTC). The investigators believe they have invested more time and effort into developing this line of investigation than any other group in the World. The investigators first reviewed the pertinent literature and subsequently retrospectively reviewed the outcomes of this entity at both this institution and with collaborators at other CTTC sites. The investigators have examined the anatomic and practical reasons as to why OPTXs are occult, as well as novel investigation methods to detect them during the initial evaluation for trauma, and documented the morbidity that may occur with their treatment.

ELIGIBILITY:
Inclusion Criteria:

1. age >= 18 years old
2. small to moderate sized occult pneumothorax identified on chest or abdominal CT scan
3. no chest drain in-situ
4. no hemothorax which warrants drainage in the judgment of attending clinician
5. no respiratory compromise in the judgment of the attending clinician

Exclusion Criteria:

1. not expected to survive
2. large occult pneumothorax
3. pneumothorax obvious on plain CXR (not occult)
4. respiratory distress in the judgment of the attending clinician
5. pre-existing chest drain in-situ

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2006-08; Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Outcome Variables: In ventilated patients with small to moderate sized occult PTXs, the rate of respiratory distress will not differ between those treated with chest thoracostomy tubes and those not treated but simply observed | admission to hospital discharge

SECONDARY OUTCOMES:
Observation of small OPTXs in ventilated patients will not increases the rates of Emergency chest drainage, Death, tracheostomy, ARDS, Ventilator associated pneumonia (VAP), or the Abdominal Compartment Syndrome (ACS) | admission to hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Andrew W Kirkpatrick, MD, Principal Investigator — Canadian Trauma Trials Collaborative
Locations (4):
- Canada (4):
  - Foothills Medical Centre, Calgary, Alberta
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Centre Hospitalier Affilie Universitaire de Quebec, Québec, Quebec
  - University of Sherbrooke, Sherbrooke

IPD SHARING:
Plan to Share IPD: No
No plan.

REFERENCES:
- [Background] Ball CG, Hameed SM, Evans D, Kortbeek JB, Kirkpatrick AW; Canadian Trauma Trials Collaborative. Occult pneumothorax in the mechanically ventilated trauma patient. Can J Surg. 2003 Oct;46(5):373-9. PMID 14577712
- [Background] Ball CG, Kirkpatrick AW, Laupland KB, Fox DL, Litvinchuk S, Dyer DM, Anderson IB, Hameed SM, Kortbeek JB, Mulloy R. Factors related to the failure of radiographic recognition of occult posttraumatic pneumothoraces. Am J Surg. 2005 May;189(5):541-6; discussion 546. doi: 10.1016/j.amjsurg.2005.01.018. PMID 15862493
- [Background] Ball CG, Kirkpatrick AW, Laupland KB, Fox DI, Nicolaou S, Anderson IB, Hameed SM, Kortbeek JB, Mulloy RR, Litvinchuk S, Boulanger BR. Incidence, risk factors, and outcomes for occult pneumothoraces in victims of major trauma. J Trauma. 2005 Oct;59(4):917-24; discussion 924-5. doi: 10.1097/01.ta.0000174663.46453.86. PMID 16374282
- [Background] Wall SD, Federle MP, Jeffrey RB, Brett CM. CT diagnosis of unsuspected pneumothorax after blunt abdominal trauma. AJR Am J Roentgenol. 1983 Nov;141(5):919-21. doi: 10.2214/ajr.141.5.919. PMID 6605061
- [Background] Rhea JT, Novelline RA, Lawrason J, Sacknoff R, Oser A. The frequency and significance of thoracic injuries detected on abdominal CT scans of multiple trauma patients. J Trauma. 1989 Apr;29(4):502-5. doi: 10.1097/00005373-198904000-00015. PMID 2709459
- [Background] Hill SL, Edmisten T, Holtzman G, Wright A. The occult pneumothorax: an increasing diagnostic entity in trauma. Am Surg. 1999 Mar;65(3):254-8. PMID 10075304
- [Background] Garramone RR Jr, Jacobs LM, Sahdev P. An objective method to measure and manage occult pneumothorax. Surg Gynecol Obstet. 1991 Oct;173(4):257-61. PMID 1925893
- [Background] Wolfman NT, Myers WS, Glauser SJ, Meredith JW, Chen MY. Validity of CT classification on management of occult pneumothorax: a prospective study. AJR Am J Roentgenol. 1998 Nov;171(5):1317-20. doi: 10.2214/ajr.171.5.9798871.
- [Background] Brasel KJ, Stafford RE, Weigelt JA, Tenquist JE, Borgstrom DC. Treatment of occult pneumothoraces from blunt trauma. J Trauma. 1999 Jun;46(6):987-90; discussion 990-1. doi: 10.1097/00005373-199906000-00001. PMID 10372613
- [Background] Neff MA, Monk JS Jr, Peters K, Nikhilesh A. Detection of occult pneumothoraces on abdominal computed tomographic scans in trauma patients. J Trauma. 2000 Aug;49(2):281-5. doi: 10.1097/00005373-200008000-00015. PMID 10963540
- [Background] Tocino IM, Miller MH, Frederick PR, Bahr AL, Thomas F. CT detection of occult pneumothorax in head trauma. AJR Am J Roentgenol. 1984 Nov;143(5):987-90. doi: 10.2214/ajr.143.5.987. PMID 6333171
- [Background] Trupka A, Waydhas C, Hallfeldt KK, Nast-Kolb D, Pfeifer KJ, Schweiberer L. Value of thoracic computed tomography in the first assessment of severely injured patients with blunt chest trauma: results of a prospective study. J Trauma. 1997 Sep;43(3):405-11; discussion 411-2. doi: 10.1097/00005373-199709000-00003. PMID 9314300
- [Background] Voggenreiter G, Aufmkolk M, Majetschak M, Assenmacher S, Waydhas C, Obertacke U, Nast-Kolb D. Efficiency of chest computed tomography in critically ill patients with multiple traumas. Crit Care Med. 2000 Apr;28(4):1033-9. doi: 10.1097/00003246-200004000-00020. PMID 10809278
- [Background] Guerrero-Lopez F, Vazquez-Mata G, Alcazar-Romero PP, Fernandez-Mondejar E, Aguayo-Hoyos E, Linde-Valverde CM. Evaluation of the utility of computed tomography in the initial assessment of the critical care patient with chest trauma. Crit Care Med. 2000 May;28(5):1370-5. doi: 10.1097/00003246-200005000-00018. PMID 10834680
- [Background] Holmes JF, Brant WE, Bogren HG, London KL, Kuppermann N. Prevalence and importance of pneumothoraces visualized on abdominal computed tomographic scan in children with blunt trauma. J Trauma. 2001 Mar;50(3):516-20. doi: 10.1097/00005373-200103000-00017. PMID 11265032
- [Background] Rowan KR, Kirkpatrick AW, Liu D, Forkheim KE, Mayo JR, Nicolaou S. Traumatic pneumothorax detection with thoracic US: correlation with chest radiography and CT--initial experience. Radiology. 2002 Oct;225(1):210-4. doi: 10.1148/radiol.2251011102. PMID 12355007
- [Background] Collins JC, Levine G, Waxman K. Occult traumatic pneumothorax: immediate tube thoracostomy versus expectant management. Am Surg. 1992 Dec;58(12):743-6. PMID 1456598
- [Background] American College of Surgeons. Advanced trauma life support course for doctors. Committee on Trauma: Instructors' Course Manual. Chicago, 1997.
- [Background] Etoch SW, Bar-Natan MF, Miller FB, Richardson JD. Tube thoracostomy. Factors related to complications. Arch Surg. 1995 May;130(5):521-5; discussion 525-6. doi: 10.1001/archsurg.1995.01430050071012. PMID 7748091
- [Background] Enderson BL, Abdalla R, Frame SB, Casey MT, Gould H, Maull KI. Tube thoracostomy for occult pneumothorax: a prospective randomized study of its use. J Trauma. 1993 Nov;35(5):726-9; discussion 729-30. PMID 8230337
- [Background] Wilson H, Ellsmere J, Talon J, Kirkpatrick A. Natural history of the occult pneumothorax in the blunt trauma patient. Journal of Trauma 59(2): 541, 2005.
- [Background] Wilson H, Ellsmere J, Tallon J, Kirkpatrick A. Occult pneumothorax in the blunt trauma patient requiring surgery: a qualitative review. Journal of Trauma 59(2): 545, 2005
- [Background] Ball CG, Kirkpatrick AW, Fox DL, Laupland KB, Louis LJ, Andrews GD, Dunlop MP, Kortbeek JB, Nicolaou S. Are occult pneumothoraces truly occult or simply missed? J Trauma. 2006 Feb;60(2):294-8 discussion 298-9. doi: 10.1097/01.ta.0000202462.96207.18. PMID 16508485
- [Background] Sargsyan AE, Hamilton DR, Nicolaou S, Kirkpatrick AW, Campbell MR, Billica RD, Dawson D, Williams DR, Melton SL, Beck G, Forkheim K, Dulchavsky SA. Ultrasound evaluation of the magnitude of pneumothorax: a new concept. Am Surg. 2001 Mar;67(3):232-5; discussion 235-6. PMID 11270880
- [Background] Kirkpatrick AW, Simons RK, Brown DR, Ng AK, Nicolaou S. Digital hand-held sonography utilised for the focused assessment with sonography for trauma: a pilot study. Ann Acad Med Singap. 2001 Nov;30(6):577-81. PMID 11817283
- [Background] Kirkpatrick AW, Ng AK, Dulchavsky SA, Lyburn I, Harris A, Torregianni W, Simons RK, Nicolaou S. Sonographic diagnosis of a pneumothorax inapparent on plain radiography: confirmation by computed tomography. J Trauma. 2001 Apr;50(4):750-2. doi: 10.1097/00005373-200104000-00029. No abstract available. PMID 11303179
- [Background] Cunningham J, Kirkpatrick AW, Nicolaou S, Liu D, Hamilton DR, Lawless B, Lee M, Brown DR, Simons RK. Enhanced recognition of "lung sliding" with power color Doppler imaging in the diagnosis of pneumothorax. J Trauma. 2002 Apr;52(4):769-71. doi: 10.1097/00005373-200204000-00029. No abstract available. PMID 11956400
- [Background] Dulchavsky SA, Schwarz KL, Kirkpatrick AW, Billica RD, Williams DR, Diebel LN, Campbell MR, Sargysan AE, Hamilton DR. Prospective evaluation of thoracic ultrasound in the detection of pneumothorax. J Trauma. 2001 Feb;50(2):201-5. doi: 10.1097/00005373-200102000-00003. PMID 11242282
- [Background] Kirkpatrick A, Nicolaou S. The sonographic detection of pneumothoraces (pages 227-234). In: Kharmy-Jones R, Nathens A, Stern E (editors). Thoracic Trauma and Critical Care. Boston: Kleuwer Academic Publishers. 2002.
- [Background] Hamilton DR, Sargsyan AE, Kirkpatrick AW, Nicolaou S, Campbell M, Dawson DL, Melton SL, Beck G, Guess T, Rasbury J, Dulchavsky SA. Sonographic detection of pneumothorax and hemothorax in microgravity. Aviat Space Environ Med. 2004 Mar;75(3):272-7. PMID 15018297
- [Background] Kirkpatrick AW, Sirois M, Laupland KB, Liu D, Rowan K, Ball CG, Hameed SM, Brown R, Simons R, Dulchavsky SA, Hamiilton DR, Nicolaou S. Hand-held thoracic sonography for detecting post-traumatic pneumothoraces: the Extended Focused Assessment with Sonography for Trauma (EFAST). J Trauma. 2004 Aug;57(2):288-95. doi: 10.1097/01.ta.0000133565.88871.e4. PMID 15345974
- [Background] Kirkpatrick AW, Nicolaou S, Rowan K, Liu D, Cunningham J, Sargsyan AE, Hamilton D, Dulchavsky SA. Thoracic sonography for pneumothorax: the clinical evaluation of an operational space medicine spin-off. Acta Astronaut. 2005 May-Jun;56(9-12):831-8. doi: 10.1016/j.actaastro.2005.01.008. PMID 15835018
- [Background] Ball CG, Lord J, Laupland KB, Gmora S, Mulloy RH, Ng AK, Schieman C, Kirkpatrick AW. Chest tube complications: how well are we training our residents? Can J Surg. 2007 Dec;50(6):450-8. PMID 18053373